CLINICAL TRIAL: NCT03252015
Title: Multiple-Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Drug-Drug Interaction Study of Lasmiditan
Brief Title: A Study of Multiple Doses of Lasmiditan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 16859; H8H-MC-LAHE (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-08-15; First posted 2017-08-16 (Actual); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Probe Drug Cocktail (Cohort 1a) (Experimental): Probe Drug Cocktail administered orally on Day -3.
  Interventions: Drug: Probe Drug Cocktail
- 200 milligrams (mg) Lasmiditan+Probe Drug Cocktail (Cohort 1) (Experimental): 200 mg lasmiditan administered alone, orally, on Days 1-6 and concurrently with probe drug cocktail on Day 7.
  Interventions: Drug: Probe Drug Cocktail; Drug: Lasmiditan
- Placebo+Probe Drug Cocktail (Cohort 1b) (Placebo Comparator): Placebo administered alone, orally, on Days 1-6 and concurrently with probe drug cocktail on Day 7.
  Interventions: Drug: Probe Drug Cocktail; Drug: Placebo
- 400 mg Lasmiditan (Cohort 2a) (Experimental): 400 mg lasmiditan administered orally for 7 days.
  Interventions: Drug: Lasmiditan
- Placebo (Cohort 2b) (Experimental): Placebo administered orally for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probe Drug Cocktail — Administered orally
  Arms: 200 milligrams (mg) Lasmiditan+Probe Drug Cocktail (Cohort 1); Placebo+Probe Drug Cocktail (Cohort 1b); Probe Drug Cocktail (Cohort 1a)
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: 200 milligrams (mg) Lasmiditan+Probe Drug Cocktail (Cohort 1); 400 mg Lasmiditan (Cohort 2a)
Drug: Placebo — Administered orally
  Arms: Placebo (Cohort 2b); Placebo+Probe Drug Cocktail (Cohort 1b)

SUMMARY:
The purpose of this study is to look at how much lasmiditan, study drug, gets into the blood stream and how long it takes the body to get rid of it.

When drugs are taken together, one or all of the drugs used in combination may be affected. This study will also evaluate the concentrations in the blood of a probe drug cocktail taken alone and in combination with lasmiditan. Information about any side effects that may occur will also be collected.

The study has two parts. Participants will only enroll in one part. This study will last about 25 days for group 1 and 22 days for group 2, not including screening. Screening is required within 28 days prior to the start of the study.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, as determined by medical history and physical examination
* Have a body mass index (BMI) of 19.0 to 35.0 kilograms per meter squared (kg/m²) inclusive, at the time of screening

Exclusion Criteria:

* Have participated, within the last 30 days, in a clinical study involving an Investigational Product (IP)
* Have previously completed or withdrawn from this study or any other study investigating Lasmiditan, and have previously received Lasmiditan
* Have clinically significant abnormality in the 12-lead ECG, including corrected QT interval (QTc) with Fridericia's correction (QTcF) greater than (>) 450 milliseconds (ms) for men or >470 ms for women or any abnormality that in the opinion of the investigator increases the risk of participating in the study (not limited to significant bradycardia or heart block)
* History of, show evidence of, or are undergoing treatment for significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression), have a recent history of a suicide attempt (30 days within screening visit and any time between screening visit and baseline); or are clinically judged by the investigator to be at risk for suicide
* History of hypoglycemia
* Known history of glucose-6-phosphate dehydrogenase deficiency
* Are taking a concomitant medication or a dietary substance that affects cytochrome P450 (CYP)1A2, CYP2C9, and/or CYP3A isotypes within 14 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Daytona Beach, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1a (Placebo+Probe Drug Cocktail): Placebo administered alone, orally (PO), on Days 1-6 and concurrently with probe drug cocktail on Day -3 and Day 7.
- Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail): Daily,oral (PO), 200 mg lasmiditan Days 1-6 and concurrently with probe drug cocktail on Days -3 and Day 7.
- Cohort 2a (Placebo): Placebo administered daily PO, Days 1-7.
- Cohort 2b (400 mg Lasmiditan): Daily,oral (PO), 400 mg lasmiditan Days 1-7
Period: Overall Study
Arm/Group | Cohort 1a (Placebo+Probe Drug Cocktail) | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail) | Cohort 2a (Placebo) | Cohort 2b (400 mg Lasmiditan)
Started | 12 | 28 | 15 | 15
Received at Least 1 Dose of Study Drug | 12 | 28 | 15 | 15
Completed | 11 | 27 | 14 | 14
Not Completed | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Cohort 1a (Placebo+Probe Drug Cocktail): Placebo administered alone, orally, on Days 1-6 and concurrently with probe drug cocktail on Day 7.
- Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail): Daily,oral (PO), 200 mg lasmiditan Days 1-6 and concurrently with probe drug cocktail on Day 7.
- Total: Total of all reporting groups
Arm/Group | Cohort 1a (Placebo+Probe Drug Cocktail) | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail) | Cohort 2a (Placebo) | Cohort 2b (400 mg Lasmiditan) | Total
Number analyzed (Participants) | 12 | 28 | 15 | 15 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (11.9) | 42.9 (12.3) | 39.5 (11.4) | 36.9 (9.7) | 40.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 6 | 6 | 30
  Male | 6 | 16 | 9 | 9 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 5 | 8 | 31
  Not Hispanic or Latino | 4 | 18 | 10 | 7 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 13 | 7 | 7 | 31
  White | 8 | 15 | 8 | 7 | 38
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 28 | 15 | 15 | 70
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 74.78 (13.14) | 81.92 (13.72) | 74.13 (11.04) | 78.95 (14.67) | 78.39 (13.45)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] | 27.17 (2.54) | 28.18 (3.51) | 25.87 (3.32) | 27.14 (3.88) | 27.29 (3.45)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module. Adverse events for this outcome measure are reported by arm. SAEs are reported by study drug in the Adverse Events module.
Time Frame: Baseline through 14 days after last administration of study drug
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a (Placebo+Probe Drug Cocktail) | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail) | Cohort 2a (Placebo) | Cohort 2b (400 mg Lasmiditan)
Number analyzed (Participants) | 12 | 28 | 15 | 15
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Lasmiditan on Day 1
Description: PK: Cmax of lasmiditan
Time Frame: Lasmiditan PK: Day 1:0.5 hour (hr), 1hr , 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, 12hr, 24hr and 48 hr postdose
Population: All participants who received at least 1 dose of lasmiditan on Day 1 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 200 mg Lasmiditan: Daily,oral (PO), 200 mg lasmiditan Days 1-6 and concurrently with probe drug cocktail on Day 7.
- 400 mg Lasmiditan: Daily,oral (PO), 400 mg lasmiditan Days 1-7
Arm/Group | 200 mg Lasmiditan | 400 mg Lasmiditan
Number analyzed (Participants) | 28 | 15
nanograms per milliliter (ng/mL) | 349 (32) | 750 (44)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Lasmiditan on Day 7
Description: PK: Cmax of lasmiditan Day 7
Time Frame: Lasmiditan PK: Day 7: 0.5hour(hr), 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, 12hr, 24hr postdose
Population: All participants who received at least 1 dose of lasmiditan on Day 7 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 200 mg Lasmiditan | 400 mg Lasmiditan
Number analyzed (Participants) | 26 | 14
ng/mL | 353 (29) | 808 (41)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve to the End of the Dosing Period (AUC[Tau]) Lasmiditan on Day 1
Description: PK: AUCtau of lasmiditan
Time Frame: Day 1:0.5 hour (hr), 1hr , 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, 12hr, and 24hr postdose
Population: All participants who received at least 1 dose of lasmiditan on Day 1 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hour per milliLiter
Arm/Group | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail) | Cohort 2b (400 mg Lasmiditan)
Number analyzed (Participants) | 28 | 15
nanograms times hour per milliLiter | 2070 (32) | 4530 (39)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve to the End of the Dosing Period (AUC[Tau]) Lasmiditan on Day 7
Description: PK AUCtau of lasmiditan
Time Frame: Lasmiditan PK: Day 7: 0.5hour(hr), 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, 12hr,and 24hr postdose
Population: All participants who received at least 1 dose of lasmiditan on Day 1 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms time hours per milliLiter
Groups:
- 200 mg Lasmiditan+Probe Drug Cocktail (Cohort 1): Daily,oral (PO), 200 mg lasmiditan Days 1-6 and concurrently with probe drug cocktail on Day 7.
- 400 mg Lasmiditan (Cohort 2): Daily,oral (PO), 400 mg lasmiditan Days 1-7
Arm/Group | 200 mg Lasmiditan+Probe Drug Cocktail (Cohort 1) | 400 mg Lasmiditan (Cohort 2)
Number analyzed (Participants) | 26 | 14
nanograms time hours per milliLiter | 2160 (29) | 4690 (36)

6. Secondary Outcome: Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ) Total Score
Description: BWSQ is a 20 item, self administered withdrawal symptom questionnaire. Each question is scored by a 0 representing no withdrawal symptoms, 1 for moderate symptoms, 2 for severe symptoms. Total score at each time point will be averaged for each treatment in each cohort.
Time Frame: PreDose Day 7 and Day 21
Population: All participants who received at least 1 dose of study drug and completed the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1a (Placebo+Probe Drug Cocktail) | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail) | Cohort 2a (Placebo) | Cohort 2b (400 mg Lasmiditan)
Number analyzed (Participants) | 12 | 28 | 15 | 15
units on a scale
  Day 7: number analyzed (Participants) | 11 | 27 | 13 | 14
  Day 7 | 0.0 (0.0) | 0.2 (0.6) | 0.0 (0.0) | 0.1 (0.3)
  Day 21: number analyzed (Participants) | 12 | 28 | 15 | 14
  Day 21 | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Cohort 1a (Placebo+Probe Drug Cocktail) vs Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail); Day 7; Test type: Superiority; Mean Difference (Final Values) = -0.182, 95% CI 2-sided [-0.412 to 0.049]
Statistical Analysis 2: Comparison: Cohort 2a (Placebo) vs Cohort 2b (400 mg Lasmiditan); Day 7; Test type: Superiority; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.081 to 0.224]
Statistical Analysis 3: Comparison: Cohort 1a (Placebo+Probe Drug Cocktail) vs Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail); Day 21; Test type: Superiority; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [0.000 to 0.000]
Statistical Analysis 4: Comparison: Cohort 2a (Placebo) vs Cohort 2b (400 mg Lasmiditan); Day 21; Test type: Superiority; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [0.000 to 0.000]

7. Secondary Outcome: Physician Withdrawal Checklist (PWC)Total Score
Description: Physician Withdrawal Checklist (PWC) : 20 item physician rated interview measuring anxiolytic drug withdrawal-related signs and symptoms (gastrointestinal, mood, sleep, motor, somatic, perception and cognition); range 0 (not present) to 3 (severe); total score range: 0 to 60; higher score = more affected.
Time Frame: Day 7 and Day 21 at anytime
Population: All participants who received at least 1 dose of study drug and had completed the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1a (Placebo+Probe Drug Cocktail) | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail) | Cohort 2a (Placebo) | Cohort 2b (400 mg Lasmiditan)
Number analyzed (Participants) | 12 | 28 | 15 | 14
units on a scale
  Day 7 Predose: number analyzed (Participants) | 11 | 27 | 13 | 14
  Day 7 Predose | 0.2 (0.4) | 0.0 (0.2) | 0.0 (0.0) | 0.1 (0.3)
  Day 21 | 0.0 (0.0) | 0.1 (0.4) | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Cohort 1a (Placebo+Probe Drug Cocktail) vs Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail); Day 7; Test type: Superiority; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.340 to 0.050]
Statistical Analysis 2: Comparison: Cohort 2a (Placebo) vs Cohort 2b (400 mg Lasmiditan); Test type: Superiority; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.081 to 0.224]
Statistical Analysis 3: Comparison: Cohort 1a (Placebo+Probe Drug Cocktail) vs Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail); Day 21; Test type: Superiority; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [-0.151 to 0.294]
Statistical Analysis 4: Comparison: Cohort 2a (Placebo) vs Cohort 2b (400 mg Lasmiditan); Day 21; Test type: Superiority; Mean Difference (Final Values) = 0.000, 95% CI 2-sided [0.000 to 0.000]

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Metabolite M8 on Day 1
Description: Cmax of M8 on Day 1 following a single and repeated oral daily dosing of 200 and 400 mg lasmiditan. M8 is a metabolite of lasmiditan.
Time Frame: Day 1: 0.5 hr, 1hr, 1.5hr, 2 hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, 12hr, 24 hr adn 48 hr postdose
Population: All participant who received at least 1 dose of lasmiditan and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/mL
Arm/Group | 200 mg Lasmiditan | 400 mg Lasmiditan
Number analyzed (Participants) | 28 | 15
mg/mL | 407 (24) | 964 (18)

9. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Metabolite M8 on Day 7
Description: Cmax of M8 on Day 7 following a single and repeated oral daily dosing of 200 and 400 mg lasmiditan. M8 is a metabolite of lasmiditan.
Time Frame: Day 7: Predose, 0.5hr, 1hr, 1.5hr, 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, 12hr, 24 hr and 48 hr postdose
Population: All participants who received at least one dose of lasmiditan and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 200 mg Lasmiditan+Probe Drug Cocktail (Cohort 1) | 400 mg Lasmiditan (Cohort 2)
Number analyzed (Participants) | 26 | 14
ng/mL | 641 (20) | 1500 (20)

10. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Midazolam
Description: PK: Cmax of midazolam.
Time Frame: Day -3: Predose, 0.5 hour(hr), 1hr, 1.5hr. 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, and 12 hr postdose,
Population: All randomized participant who received midazolam on Day -3 and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliLiter
Groups:
- Participants Who Received Probe Drug Cocktail: Probe drug cocktail was administered PO alone to all participants on Day -3.
Arm/Group | Participants Who Received Probe Drug Cocktail
Number analyzed (Participants) | 40
nanograms per milliLiter | 10. (39)

11. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Midazolam on Day 7
Description: PK of midazolam.
Time Frame: Day 7:Predose, 0,5hr,1hr, 1.5hr. 2hr, 2.5hr, 3hr, 4hr, 6hr, 8hr, and 12 hr postdose
Population: All randomized participant who received midazolam on Day 7 and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Cohort 1a (Placebo+Probe Drug Cocktail) | Cohort 1b (200 mg Lasmiditan+Probe Drug Cocktail)
Number analyzed (Participants) | 11 | 27
nanograms per milliliter | 10.1 (40) | 9.45 (34)

ADVERSE EVENTS:
Time Frame: Baseline through 28 days
Description: All participants who received at least 1 dose of study drug.
Groups:
- Probe Drug Cocktail (Cohort 1): Probe drug cocktail administered on Day 13 and Day 7
- 200 mg Lasmiditan QD (Cohort 1): Daily,oral (PO), 200 mg lasmiditan Days 1-6
- 200 mg Lasmiditan QD + Probe Drug Cocktail (Cohort 1): Daily,oral (PO), 200 mg lasmiditan Days 1-6 and concurrently with probe drug cocktail on Day 7.
- Placebo QD (Cohort 1); Placebo QD (Cohort 2): Placebo administered daily PO, Days 1-7
- Placebo QD + Probe Drug Cocktail (Cohort 1): Placebo administered alone, orally (PO), on Days 1-6 and concurrently with probe drug cocktail on Day -3 and Day 7
- 400 mg Lasmiditan QD (Cohort 2): Daily,oral (PO), 400 mg lasmiditan Days 1-7
Arm/Group | Probe Drug Cocktail (Cohort 1) | 200 mg Lasmiditan QD (Cohort 1) | 200 mg Lasmiditan QD + Probe Drug Cocktail (Cohort 1) | Placebo QD (Cohort 1) | Placebo QD + Probe Drug Cocktail (Cohort 1) | 400 mg Lasmiditan QD (Cohort 2) | Placebo QD (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/28 | 0/27 | 0/12 | 0/11 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/28 | 0/27 | 0/12 | 0/11 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/40 | 13/28 | 4/27 | 5/12 | 1/11 | 5/15 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probe Drug Cocktail (Cohort 1) (N=40) | 200 mg Lasmiditan QD (Cohort 1) (N=28) | 200 mg Lasmiditan QD + Probe Drug Cocktail (Cohort 1) (N=27) | Placebo QD (Cohort 1) (N=12) | Placebo QD + Probe Drug Cocktail (Cohort 1) (N=11) | 400 mg Lasmiditan QD (Cohort 2) (N=15) | Placebo QD (Cohort 2) (N=15)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrong technique in product usage process (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 6 (8) | 2 (2) | 0 (0) | 0 (0) | 3 (7) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT03252015/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT03252015/SAP_001.pdf